CLINICAL TRIAL: NCT03286127
Title: Assessment of Palliative Care in Inpatient and Outpatient Settings Using the Integrated Palliative Care Outcome Scale: a Multi-centric Observational Study
Brief Title: Palliative Outcome Evaluation Muenster I
Acronym: POEM I
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Muenster (Other)
Collaborators: St. Franziskus Hospital (Other); Raphaelsklinik Münster (Unknown); Josephs Hospital Warendorf (Unknown); Palliativnetz Muenster gGmbH (Unknown)
Responsible Party: Sponsor
Other Study IDs: UKM_POEM I
Record Dates: First submitted 2017-09-14; First posted 2017-09-18 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Cancer; Chronic Heart Failure; COPD Exacerbation; Palliative Care
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- PCU (unit): Those patients who received specialised palliative care on a palliative care unit.(palliative care unit)
  Interventions: Other: specialized palliative care
- IPCC (hospital): Those patients admitted to a regular hospital ward who received specialised palliative care from an inpatient palliative care consultation team.
  (inpatient palliative care consultation team)
  Interventions: Other: specialized palliative care
- OPCC (outpatient): Those patients who received specialised palliative care at home from an outpatient palliative care consultation team. (outpatient palliative care consultation team)
  Interventions: Other: specialized palliative care

INTERVENTIONS:
Other: specialized palliative care — specialized palliative care provided in different settings

SUMMARY:
For patients with an advanced disease and their families an excellent and compassionate care is essential. However, in hospitals optimal end-of-life care is not yet fully realized and patient's needs are often not met. Palliative care is able to increase patients' quality of life and to carefully meet their and their families' needs.

To improve the awareness of unmet needs patient-reported outcome measurement has been the pivot of latest palliative care research. Besides the improvement of care outcome measurement allows the evaluation of the quality of palliative care and comparisons on a national and international level.

The aim of the present study is to evaluate the quality of palliative care in different settings (palliative care unit, inpatient and outpatient consultation teams) using the Integrated Palliative Care Outcome Scale (IPOS). The IPOS has been lately developed as improved follow-up version of the Palliative Care Outcome Scale (POS) integrating most important questions and simultaneously being brief and comprehensive. The study is planned as a multi-centric observational study. Primary endpoint is the reduction of symptom burden of patients.

The clinical study hypothesis bases on the assumption that palliative care can change the symptom burden, measured by a change in the IPOS overall profile score, and that there might be a difference in the size of the effect depending on the caring setting.

DETAILED DESCRIPTION:
After the enrolment and consent of participation the patient receive a questionnaire consisting of three independent assessments: To assess the symptom burden and specific palliative care needs the Integrated Palliative Outcome Scale (IPOS) is used. To measure the generic health-related quality of life the patient has to answer the EuroQoL Group 5-Dimension 5-Level Self Report Questionnaire (EQ-5D-5L). To get an opinion of the general condition the patient is to complete the NCCN Distress Thermometer which includes a visual analogue scale (with values from 0 to 10).

Meanwhile, a professional palliative caregiver completes a questionnaire about the main demographic aspects of the patients and assess the palliative care needs and the symptom burden using the IPOS.

After one week both, patient and professional palliative caregiver, will receive the same questionnaires again to assess the change from baseline.

ELIGIBILITY:
Inclusion Criteria:

* Indication for palliative care due to any advanced life-limiting and progressive disease
* 18 years and older

Exclusion Criteria:

* Age under 18 years
* pregnant or breastfeeding women
* Inability to understand information for participation
* Refusal of participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients with an advanced life-limiting and progressive disease needing palliative care. The three groups are formed depending of the setting in which palliative care will be provided.
Sampling Method: Non-Probability Sample
Enrollment: 347 (Estimated)
Dates: Start 2017-09-11 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
symptom burden (IPOS) | From Baseline to End of Follow-Up (0, 1 week)
  Change from baseline in palliative care needs and specific symptoms (at day 7) assessed with the Integrated Palliative Care Outcome Scale (IPOS). The IPOS includes 10 symptoms and 7 questions on patients and carers emotional situation, spiritual concerns, and provision of information and support. The overall profile score is the sum of the scores from each of the 17 questions.

SECONDARY OUTCOMES:
Generic health-related quality of life (EQ-5D-5L) | From Baseline to End of Follow-Up (0, 1 week)
  Change from baseline in patients' generic health-related quality of life measured with the EuroQoL Group 5-Dimension 5-Level Self Report Questionnaire (EQ-5D-5L). The EQ-5D-5L essentially consists of 2 pages - the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression). Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The visual analogue scale of the EQ-5D-5L questionnaire ranges from 0 to 100 (with 0 representing the worst health the patient can imagine and 100 representing the best health the patient can imagine).

CONTACTS AND LOCATIONS:
Locations (5):
- Germany (5):
  - Hospital St. Raphael Muenster, Münster, North Rhine-Westphalia
  - Hospital St. Franziskus Muenster, Münster, North Rhine-Westphalia
  - University Hospital Muenster, Münster, North Rhine-Westphalia
  - Palliativnetz Muenster, Münster, North Rhine-Westphalia
  - Hospital St. Josef Warendorf, Warendorf, North Rhine-Westphalia

IPD SHARING:
Plan to Share IPD: No